CLINICAL TRIAL: NCT06964945
Title: Auricular Acupressure for the Prevention of Sleep Disorder in Breast Cancer Patients: A Randomized Controlled Trial
Brief Title: Auricular Acupressure for Sleep Disorder Prevention in Breast Cancer
Acronym: AA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202500593B0; KH20250422001 (Other: Kaohsiung Chang Gung Memorial Hospital, Taiwan)
Record Dates: First submitted 2025-05-07; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Sleep Disorders Sleep Disturbance Insomnia
Keywords: Auricular acupressure, Breast cancer, Sleep disturbance
MeSH Terms: conditions — Breast Neoplasms; Parasomnias

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to either the auricular acupressure group or the sham control group using stratified block randomization based on hormone receptor status and menopausal status. Each participant receives only one type of intervention throughout the 12-week period.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors are blinded to group allocation. Randomization was performed using stratified block randomization by an independent statistician. Identical adhesive patches were used in both groups to maintain participant blinding. Outcome assessors were not involved in the intervention procedures and were unaware of participant group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular Acupressure (AA) (Experimental): Participants in this group receive auricular acupressure using Vaccaria seeds applied to five specific auricular acupoints over 12 weeks. All participants also receive standard sleep hygiene education.
  Interventions: Behavioral: Auricular Acupressure with Vaccaria Seeds
- Sham Auricular Acupressure (Sham Comparator): Participants in this group receive sham auricular acupressure using identical adhesive patches without Vaccaria seeds applied to the same five auricular acupoints. The procedure mimics the true intervention in appearance, duration, and frequency, maintaining participant blinding. All participants also receive standardized sleep hygiene education.
  Interventions: Behavioral: Sham Auricular Acupressure (No Seeds)

INTERVENTIONS:
Behavioral: Auricular Acupressure with Vaccaria Seeds — Auricular Acupressure with Vaccaria Seeds Participants in this group receive auricular acupressure using 2 mm Vaccaria seeds adhered to five specific auricular acupoints (TF4, CO15, Extra5, LO4, LO4) with 7 mm × 7 mm adhesive patches. Each session lasts 10-20 minutes, with seeds left in place for 5-7 days. A total of 12 weeks, along with standardized sleep hygiene education.
  Arms: Auricular Acupressure (AA)
Behavioral: Sham Auricular Acupressure (No Seeds) — Participants in this group receive sham auricular acupressure using identical adhesive patches without Vaccaria seeds, applied to the same five auricular points. Procedures, duration, frequency, and sleep hygiene education are identical to those in the experimental group to maintain blinding.
  Arms: Sham Auricular Acupressure

SUMMARY:
Abstract

Background:

Sleep disturbances are highly prevalent among breast cancer (BC) patients, especially during chemotherapy, significantly affecting quality of life and treatment adherence. Conventional pharmacologic treatments for sleep disorders may cause side effects and are not always effective. Auricular acupressure (AA), a non-invasive alternative therapy, has demonstrated promising effects on sleep improvement. However, high-quality evidence for its use in BC patients remains limited.

Objective:

This study aims to evaluate the effectiveness of auricular acupressure in preventing sleep disturbances in breast cancer patients undergoing chemotherapy.

Methods:

This double-blind, randomized, sham-controlled trial will recruit 128 participants diagnosed with stage I-III breast cancer who are undergoing chemotherapy or hormone therapy. Eligible participants will be randomly assigned in a 1:1 ratio to receive either auricular acupressure (AA) or sham AA, in addition to usual care. The intervention will be administered over a 12-week period, followed by a 4-week follow-up.

In the AA group, Vaccaria seeds will be applied to five specific auricular acupoints. In the sham AA group, identical adhesive patches without seeds will be applied to the same acupoints. Both groups will receive the same treatment schedule and standardized care instructions to ensure blinding.

The primary outcome is sleep quality, assessed using the Pittsburgh Sleep Quality Index (PSQI) at baseline, and at weeks 4, 8, 12, and 16. Secondary outcomes include fatigue (measured by the BFI-T), anxiety and depression (measured by the HADS), and hypnotic medication use, assessed at baseline, and at weeks 4, 8, and 12.

Statistical analysis will be performed using Generalized Estimating Equations (GEE) to examine changes over time and between groups.

Expected Results:

We hypothesize that AA will significantly improve sleep quality and reduce symptom burden compared to sham AA in BC patients.

Conclusion:

This study will provide rigorous evidence on the efficacy and safety of auricular acupressure as a complementary intervention for sleep disturbance prevention in breast cancer patients receiving chemotherapy.

DETAILED DESCRIPTION:
Breast cancer (BC) patients frequently experience sleep disturbances throughout the treatment continuum, with prevalence rates as high as 60-87%. These disturbances are associated with increased physical and psychological burden, impaired treatment adherence, and reduced quality of life. Chemotherapy and hormone therapy, particularly those involving corticosteroids such as dexamethasone, have been identified as major contributors to sleep disruption. Although pharmacological approaches are commonly used to manage sleep issues, they are often accompanied by side effects and limited long-term efficacy.

Auricular acupressure (AA), a non-invasive technique derived from Traditional Chinese Medicine, involves stimulating specific ear points using Vaccaria seeds to regulate neurohumoral function. Previous studies have demonstrated its effectiveness in general populations with insomnia, but rigorous evidence supporting its role in cancer-related sleep disturbance-especially among BC patients-remains limited.

This double-blind, randomized, sham-controlled trial aims to evaluate the effectiveness of AA in preventing sleep disturbances in BC patients undergoing chemotherapy or hormone therapy. A total of 128 participants with stage I-III BC and no pre-existing sleep disorders will be randomized in a 1:1 ratio to receive either AA or sham AA over a 12-week period. Vaccaria seeds will be applied to five auricular points in the intervention group, while identical patches without seeds will be used in the sham group. Both groups will receive standardized sleep hygiene education.

The primary outcome is sleep quality, assessed using the Pittsburgh Sleep Quality Index (PSQI). Secondary outcomes include fatigue (BFI-T), anxiety and depression (HADS), and hypnotic medication use. Assessments will be conducted at baseline and during follow-up at weeks 4, 8, 12, and 16. Statistical analysis will use Generalized Estimating Equations (GEE) to compare changes over time between groups.

This study is expected to provide high-quality evidence on the use of AA as a complementary strategy for sleep disturbance prevention in BC patients, addressing a critical yet under-recognized aspect of supportive cancer care.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18 years or older

Histologically confirmed stage I-III breast cancer

Scheduled to undergo at least four cycles of adjuvant or neoadjuvant chemotherapy or currently receiving hormone therapy

Pittsburgh Sleep Quality Index (PSQI) score < 5 at baseline (indicating no pre-existing sleep disorder)

Able to provide informed consent and comply with study procedures

Exclusion Criteria:

* Pregnant or breastfeeding

Diagnosed with stage IIIB, inflammatory, or metastatic breast cancer

Pre-existing anemia or hematologic disorders

History of alcohol or substance abuse

Diagnosed endocrine disorders or other medical conditions affecting sleep

Active psychiatric disorders interfering with participation

Skin lesions, infections, or allergy to adhesive patches on both ears

Currently undergoing other complementary sleep-related therapies (e.g., aromatherapy, massage, herbal medicine, health supplements)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep disturbance assessed by PSQI | Baseline, Week 4, Week 8, Week 12, and follow-up at Week 16
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), a validated 19-item self-report questionnaire.

SECONDARY OUTCOMES:
Fatigue Severity Assessed by BFI-T | Baseline, Week 4, Week 8, Week 12
  Fatigue will be assessed using the Brief Fatigue Inventory - Traditional Chinese version (BFI-T), a 9-item self-report scale measuring fatigue severity and interference. Scores range from 0 (no fatigue) to 10 (severe fatigue).
Anxiety and Depression (assessed by HADS) | Baseline, Week 4, Week 8, Week 12
  Emotional distress will be measured using the Hospital Anxiety and Depression Scale (HADS), consisting of two subscales: HADS-A for anxiety and HADS-D for depression. Each subscale includes 7 items scored from 0 to 21.
Hypnotic Medication Use | Week 4, Week 8, Week 12
  Participants will record daily use of hypnotic medications, including benzodiazepines, non-benzodiazepines, antidepressants, melatonin receptor agonists, and other sleep aids. Data will be summarized as weekly usage scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data including demographic variables (e.g., age, menopausal status), group assignment (intervention vs. control), and outcome measures such as PSQI scores, BFI-T scores, HADS scores, and hypnotic medication use will be shared.
Supporting Information: Study Protocol, SAP